CLINICAL TRIAL: NCT06070610
Title: The Effect of Multiple Oral Doses of BI 1015550 on the Pharmacokinetics of Nintedanib and Pirfenidone Administered Single Dose to Healthy Male Subjects (Open-label, Two-period, Fixed-sequence Crossover Trial)
Brief Title: A Study in Healthy Men to Test Whether BI 1015550 Influences the Amount of Nintedanib and Pirfenidone in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0034; 2023-505522-34-00 (Registry Identifier: CTIS); U1111-1292-0376 (Registry Identifier: WHO registry)
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550; nintedanib; pirfenidone

STUDY DESIGN:
Intervention Model Description: Patients cross over from test treatment (T) to reference treatment (R) (two periods, fixed sequence).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reference treatment/Test treatment (Experimental): In the reference (R) treatment (period 1, two days of treatment), a single dose of 267 mg pirfenidone was administered on Day 1 and a single dose of 100 mg nintedanib on Day 2.
  In the test (T) treatment (period 2, ten days of treatment), 18 mg nerandomilast were administered twice daily for 10 days (Day -6 to Day 4). A single dose of 267 mg pirfenidone was administered on Day 1 and a single dose of 100 mg nintedanib was administered on Day 2.
  A washout period of at least 72 hours separated the last drug administration in the reference period from the first drug administration in the test period.
  Interventions: Drug: BI 1015550; Drug: Nintedanib; Drug: Pirfenidone

INTERVENTIONS:
Drug: BI 1015550 — BI 1015550
  Other Names: Nerandomilast; JASCAYD®
Drug: Nintedanib — Soft capsules
  Other Names: Ofev®
Drug: Pirfenidone — Film-coated tablets
  Other Names: Esbriet®

SUMMARY:
The main objective of this trial is to investigate the induction effect of multiple oral doses of BI 1015550 on the pharmacokinetics of nintedanib or pirfenidone.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders (including severe renal or hepatic impairment)
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open-label, two-period, fixed-sequence crossover trial to investigate the effect of multiple oral doses of 18 mg nerandomilast on the pharmacokinetics of single oral doses of 100 mg nintedanib or 267 mg pirfenidone.
Pre-assignment Details: 14 participants who met the inclusion and none of the exclusion criteria were included in the study. All 14 participants were treated in period 1. One of the 14 participants was discontinued after period 1 due to an adverse event. 13 participants were treated in period 2 and 1 of these subjects discontinue participation due to on-treatment adverse events. All 14 subjects completed the planned trial assessments. Participants were free to withdraw from the clinical trial at any time.
Period: Period 1 (Reference treatment period)
Arm/Group | Reference treatment/Test treatment
Started | 14
Completed | 14
Not Completed | 0
Period: Washout period
Arm/Group | Reference treatment/Test treatment
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1
Period: Period 2 (Test treatment period)
Arm/Group | Reference treatment/Test treatment
Started | 13
Completed | 12
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least 1 dose of trial drug.
Arm/Group | Reference Treatment/Test Treatment
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Pirfenidone in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of pirfenidone in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Geometric least squares mean (adjusted geometric mean) and the standard error (actually adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: At 0, 0:30, 1, 1:30, 2, 3, 4, 6, 8, 10, 12, 24 hours from pirfenidone administration (Period 1) and at 0, 0.30, 1, 1:30, 2, 3, 4, 6, 8, 10, 12, 24 hours from nerandomilast and pirfenidone administration (Period 2)
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided data for at least 1 primary PK endpoint and who were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was to be included in the PKS, even if he contributed only 1 PK parameter value for 1 period to the statistical assessment.
  Only participants with available data were included in the analysis.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanogram / milliliter (h*ng/mL)
Groups:
- Pirfenidone/Nintedanib alone (Reference): In the reference (R) treatment (period 1, two days of treatment), a single dose of 267 mg pirfenidone was administered on Day 1 and a single dose of 100 mg nintedanib on Day 2.
- Pirfenidone/Nintedanib in combination with Nerandomilast (Test): In the test (T) treatment (period 2, ten days of treatment), 18 mg nerandomilast was administered twice daily for 10 days (Day -6 to Day 4). A single dose of 267 mg pirfenidone was administered on Day 1 and a single dose of 100 mg nintedanib was administered on Day 2.
Arm/Group | Pirfenidone/Nintedanib alone (Reference) | Pirfenidone/Nintedanib in combination with Nerandomilast (Test)
Number analyzed (Participants) | 14 | 13
hour * nanogram / milliliter (h*ng/mL) | 9597.74 (NA) — Adjusted geometric standard error = 1.10 | 9786.78 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Pirfenidone/Nintedanib alone (Reference) vs Pirfenidone/Nintedanib in combination with Nerandomilast (Test); Test type: Other — Ratio of adjusted geometric means was calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model; Adjusted geometric mean ratio (%) = 101.97, 90% CI 2-sided [93.59 to 111.10] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 12.3

2. Primary Outcome: Area Under the Concentration-time Curve of Pirfenidone in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of pirfenidone in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Geometric least squares mean (adjusted geometric mean) and the standard error (actually adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanogram / milliliter (h*ng/mL)
Arm/Group | Pirfenidone/Nintedanib alone (Reference) | Pirfenidone/Nintedanib in combination with Nerandomilast (Test)
Number analyzed (Participants) | 14 | 13
hour * nanogram / milliliter (h*ng/mL) | 10146.47 (NA) — Adjusted geometric standard error = 1.09 | 10279.17 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Pirfenidone/Nintedanib alone (Reference) vs Pirfenidone/Nintedanib in combination with Nerandomilast (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 101.31, 90% CI 2-sided [93.60 to 109.65] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 11.4

3. Primary Outcome: Maximum Measured Concentration of Pirfenidone in Plasma (Cmax)
Description: Maximum measured concentration of pirfenidone in plasma (Cmax). Geometric least squares mean (adjusted geometric mean) and the standard error (actually adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanogram / milliliter (ng/mL)
Arm/Group | Pirfenidone/Nintedanib alone (Reference) | Pirfenidone/Nintedanib in combination with Nerandomilast (Test)
Number analyzed (Participants) | 14 | 13
nanogram / milliliter (ng/mL) | 2451.85 (NA) — Adjusted geometric standard error = 1.08 | 2479.00 (NA) — Adjusted geometric standard error = 1.08
Statistical Analysis 1: Comparison: Pirfenidone/Nintedanib alone (Reference) vs Pirfenidone/Nintedanib in combination with Nerandomilast (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 101.11, 90% CI 2-sided [87.36 to 117.02] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 21.4

4. Primary Outcome: Area Under the Concentration-time Curve of Nintedanib in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of nintedanib in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Geometric least squares mean (adjusted geometric mean) and the standard error (actually adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: At 24, 24:30, 25, 25:30, 26, 27, 28, 30, 32, 34, 36, 48, 60,72, 96 hours from pirfenidone administration (Period 1) and at 24, 24:30, 25, 25:30, 26, 27, 28, 30, 32, 34, 36, 48, 60,72, 96 hours from nerandomilast and pirfenidone administration (Period 2)
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanogram / milliliter (h*ng/mL)
Arm/Group | Pirfenidone/Nintedanib alone (Reference) | Pirfenidone/Nintedanib in combination with Nerandomilast (Test)
Number analyzed (Participants) | 14 | 12
hour * nanogram / milliliter (h*ng/mL) | 137.88 (NA) — Adjusted geometric standard error = 1.11 | 149.43 (NA) — Adjusted geometric standard error = 1.11
Statistical Analysis 1: Comparison: Pirfenidone/Nintedanib alone (Reference) vs Pirfenidone/Nintedanib in combination with Nerandomilast (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 108.37, 90% CI 2-sided [102.58 to 114.49] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 7.5

5. Primary Outcome: Area Under the Concentration-time Curve of Nintedanib in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of nintedanib in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Geometric least squares mean (adjusted geometric mean) and the standard error (actually adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * nanogram / milliliter (h*ng/mL)
Arm/Group | Pirfenidone/Nintedanib alone (Reference) | Pirfenidone/Nintedanib in combination with Nerandomilast (Test)
Number analyzed (Participants) | 14 | 11
hour * nanogram / milliliter (h*ng/mL) | 145.03 (NA) — Adjusted geometric standard error = 1.11 | 157.82 (NA) — Adjusted geometric standard error = 1.11
Statistical Analysis 1: Comparison: Pirfenidone/Nintedanib alone (Reference) vs Pirfenidone/Nintedanib in combination with Nerandomilast (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 108.82, 90% CI 2-sided [102.54 to 115.49] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 7.7

6. Primary Outcome: Maximum Measured Concentration of Nintedanib in Plasma (Cmax)
Description: Maximum measured concentration of nintedanib in plasma (Cmax). Geometric least squares mean (adjusted geometric mean) and the standard error (actually adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanogram / milliliter (ng/mL)
Arm/Group | Pirfenidone/Nintedanib alone (Reference) | Pirfenidone/Nintedanib in combination with Nerandomilast (Test)
Number analyzed (Participants) | 14 | 12
nanogram / milliliter (ng/mL) | 16.18 (NA) — Adjusted geometric standard error = 1.12 | 14.12 (NA) — Adjusted geometric standard error = 1.13
Statistical Analysis 1: Comparison: Pirfenidone/Nintedanib alone (Reference) vs Pirfenidone/Nintedanib in combination with Nerandomilast (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 87.24, 90% CI 2-sided [75.27 to 101.11] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 20.5

ADVERSE EVENTS:
Time Frame: - For pirfenidone and for nerandomilast + pirfenidone: From administration of pirfenidone + Residual Effect Period (REP) of 12 hours, up to 1 day - For nintedanib and for nerandomilast + nintedanib: From administration of nintedanib + REP of 3 days, up to 3 days - For nerandomilast: up to 12 days - All cause-mortality: up to 25 days
Description: Treated set (TS): The treated set included all subjects who were treated with at least 1 dose of trial drug. The treated set was used for safety analyses.
Groups:
- Pirfenidone: A single dose of 267 mg film-coated tablet of pirfenidone was administered orally on Day 1 in the reference (R) treatment period 1.
- Nintedanib: A single dose of 100 mg soft capsule of nintedanib was administered orally on Day 2 in the reference (R) treatment period 1.
- Nerandomilast: One film-coated tablet of 18 mg nerandomilast (BI 1015550) was administered orally twice daily for 8 days (Day -6 to Day -1 and Day 3 to Day 4) in the test (T) treatment period 2.
- Nerandomilast+pirfenidone: One film-coated tablet of 18 mg nerandomilast (BI 1015550) was administered orally twice daily together with a single dose of 267 mg pirfenidone on Day 1 in the test (T) treatment period 2.
- Nerandomilast+nintedanib: One film-coated tablet of 18 mg nerandomilast (BI 1015550) was administered orally twice daily together with a single dose of 100 mg nintedanib on Day 2 in the test (T) treatment period 2.
Arm/Group | Pirfenidone | Nintedanib | Nerandomilast | Nerandomilast+pirfenidone | Nerandomilast+nintedanib
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/14 | 4/14 | 3/13 | 1/13 | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=14) | Nintedanib (N=14) | Nerandomilast (N=13) | Nerandomilast+pirfenidone (N=13) | Nerandomilast+nintedanib (N=13)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 3
Headache (Nervous system disorders) | 0 | 2 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT06070610/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT06070610/SAP_001.pdf